CLINICAL TRIAL: NCT01715155
Title: A Retrospective Cohort Study on Therapeutic Management of Metastatic Breast Cancer in Clinical Practice in Bulgaria
Brief Title: Management of Metastatic Breast Cancer in Clinical Practice - Retrospective Study
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-OBG-XXX-2012/1
Record Dates: First submitted 2012-10-22; First posted 2012-10-26 (Estimated); Last update posted 2013-08-22 (Estimated); Status verified 2013-08

CONDITIONS: Metastatic Breast Cancer
Keywords: Metastatic Breast Cancer,; retrospective study,; disease progression,; clinical management
MeSH Terms: conditions — Breast Neoplasms; Disease Progression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Female patients diagnosed with metastatic breast cancer: Patients newly diagnosed with metastatic breast cancer, either De Novo or having progressed from a non-metastatic stage.

SUMMARY:
The purpose of this study is to evaluate the incidence rate of progression of disease, to describe the diagnostic and clinical management in patients with Metastatic Breast Cancer in the clinical practice in Bulgaria.

DETAILED DESCRIPTION:
A Retrospective Cohort Study on Therapeutic Management of Metastatic Breast Cancer in Clinical Practice in Bulgaria

ELIGIBILITY:
Inclusion Criteria:

* New diagnosis of breast cancer according to ICD-10 with confirmed metastasis
* Confirmed diagnosis between 1st July 2010 and 30th June 2011.
* Female patient managed for her disease at the same setting where final diagnosis of MBC was performed.

Exclusion Criteria:

* History of concurrent or other primary malignancies (except curatively resected non-melanoma skin cancer or in situ cervical cancer).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients newly diagnosed with breast cancer (according to ICD-10) with confirmed metastasis, regardless of being de novo diagnosed or progressed from a non-metastatic stage.
Sampling Method: Probability Sample
Enrollment: 171 (Actual)
Dates: Start 2012-12; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Number of progression events on a per patient-year-basis | Up to 2 years 5 months

SECONDARY OUTCOMES:
Proportion of patients among study population who have not progressed at 12 and 18 months after they were diagnosed | Up to 2 years 5 months
Median and mean time interval that elapsed between diagnosis and first objective tumor progression (TTP) event and subsequent events | Up to 2 years 5 months
Median and mean time from the date of diagnosis to the date of breast cancer progression or death whichever occurred first | Up to 2 years 5 months

CONTACTS AND LOCATIONS:
Locations (6):
- Bulgaria (6):
  - Research Site, Pleven
  - Research Site, Plovdiv
  - Research Site, Rousse
  - Research Site, Sofia
  - Research Site, Stara Zagora
  - Reaseach Site, Varna